CLINICAL TRIAL: NCT05669911
Title: Pilot Study: Evaluation of a Novel Self-Collection Device for Cervical Cancer Screening
Brief Title: Development of a Self-collection Device for Cervical Cancer Screening
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Teal Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: TLH-ED-004
Record Dates: First submitted 2022-11-08; First posted 2023-01-03 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Human Papilloma Virus Infection Type 16; Human Papilloma Virus Infection Type 18; Human Papilloma Virus
Keywords: cervical cancer screening; high risk HPV; hrHPV

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Teal Health Self-Collection Device Group (Experimental): This group will use the Teal Health Self-Collection Device to evaluate the instructions for use, usability, and satisfaction with the self-collection device. Participants will also undergo a Pap smear performed by a clinician. Self-collected and clinician-collected research samples will undergo HPV testing and cytological analysis using tests that are FDA-approved for use for HPV and Pap cytology.
  Interventions: Device: Teal Health Self-Collection Device Group

INTERVENTIONS:
Device: Teal Health Self-Collection Device Group — Participants will use the Instructions for Use to perform self-collection of cervicovaginal cells using the Teal Health Self-Collection Device, and will fill out a usability survey and a satisfaction and needs survey. A Pap smear will be performed by a clinician before or after self-collection.

SUMMARY:
Evaluation of a novel self-collection device for cervical cancer screening.

DETAILED DESCRIPTION:
The purpose of this study is to collect design and user input on the safety and effectiveness of the Teal Health self-collection device for patient self-collection of cervicovaginal samples for use with FDA-approved in vitro diagnostics indicated for high risk Human Papillomavirus (hrHPV) screening.

ELIGIBILITY:
Inclusion Criteria:

Group 1: Inclusion Criteria - General Population Group

1. Subject is 25 to 65 years of age and willing to provide informed consent.
2. Subject with intact cervix.

Group 2: Inclusion Criteria - HPV positive Population Group (HPV+ Enriched Group)

1. Subject is 25 to 65 years of age and willing to provide informed consent.
2. Subject with intact cervix.
3. Prior diagnosis of high risk HPV and/or positive cytology and/or presenting for colposcopy.

Exclusion Criteria:

1. Subject who reports current menstruation.
2. Subject is pregnant (based on self-reporting).
3. Subject has impaired decision-making capacity or unable to provide informed consent.
4. Subject is participating in another clinical study for an investigational device, drug, or biologic that, in the investigator's opinion, would interfere with the results of this study.
5. Subject has undergone partial or complete hysterectomy including removal of the cervix.
6. Subject has applied any chemical compounds to the cervical area within the 24-hours prior to study sample collection, including iodine, spermicide, douche, anti-fungal medications, generally, and specifically: Replens vaginal moisturizer and RepHresh vaginal hygiene products.
7. Subject on whom any form of cervical tissue alteration or surgery has been performed within the prior year, including: conization, Loop electrosurgical excision procedure (LEEP), laser surgery, or cryosurgery.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 235 (Actual)
Dates: Start 2022-08-28 (Actual); Primary Completion 2023-11-06 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Safety: SAEs | Acute - immediately after self-collection procedure
  Evaluate SAEs to confirm that SAEs from self-collection are equivalent to the rate of SAEs from health care provider-collection
Primary Effectiveness: Positive Percent Agreement (PPA) and Negative Percent Agreement (NPA) | Up to 30 days
  Detection of high risk HPV in self-collected as compared to clinician-collected sample results.
Primary Effectiveness: Sample Inadequacy Rate | Up to 30 days
  Sample inadequacy rate defined as percent of high risk HPV DNA concentrations below the detection thresholds as determined by the manufacturer.

SECONDARY OUTCOMES:
Usability Survey | Immediately After Self-collection Procedure
  Usability Survey data will be analyzed to determine device design issues (There is no scale - questions are assessed individually)
Satisfaction and Needs Survey | Immediately After Self-collection Procedure
  Satisfaction and Needs Survey data will be used to assess subjects' general willingness to use an HPV self-collection device, and concerns about HPV self-collection. (There is no scale - questions are assessed individually)
Rate of sample adequacy for liquid-based cytology analysis | Up to 30 days
  Samples will be assessed to determine if there is an adequate number of cells for liquid-based cytology analysis

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Crescendo MD, Portola Valley, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Woman's Hospital, Baton Rouge, Louisiana
  - Boston Metro, Westwood, Massachusetts
  - Planned Parenthood Gulf Coast, Houston, Texas
  - University of Wisconsin - Madison, Madison, Wisconsin